CLINICAL TRIAL: NCT05746338
Title: Validation of a Ring-type Wearable Device for Blood Oxygen Monitoring and Obstructive Sleep Apnea Syndrome Screening in Adult Chinese
Brief Title: Validation of a Ring-type Wearable Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension and the Department of Hypertension, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RING
Record Dates: First submitted 2023-01-31; First posted 2023-02-27 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea syndrome; Blood oxygen saturation; Ring-type wearable device; Polysomnography; Validation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ring-type wearable device (Experimental): The ring-type wearable device achieved continuous monitoring of blood oxygen saturation during sleep and established a OSAS screening algorithm based on oxygen saturation, which might become a complement to polysomnography.
  Interventions: Device: Ring-type wearable device
- Polysomnography (Active Comparator): Overnight polysomnography (PSG) monitor was used as the gold standard to: 1) examine the accuracy of blood oxygen monitoring assessed via a ring-type wearable device in comparison to traditional finger clip pulse oximeter; 2) assess the agreement between the ring-type wearable device and PSG monitor on OSAS screening.
  Interventions: Device: Overnight polysomnography

INTERVENTIONS:
Device: Ring-type wearable device — The ring-type wearable device is a slim, lightweight smart ring that continuously tracks blood oxygen saturation and heart rate throughout the day.
  Other Names: RingConn Smart Ring
  Arms: Ring-type wearable device
Device: Overnight polysomnography — Overnight polysomnography is the gold standard for diagnosing OSAS.
  Other Names: PSG
  Arms: Polysomnography

SUMMARY:
Study name: Validation of a Ring-type Wearable Device for Blood Oxygen Monitoring and Obstructive Sleep Apnea Syndrome Screening in Adult Chinese.

Objective: 1) To examine the accuracy of blood oxygen monitoring assessed via a ring-type wearable device in comparison to traditional finger clip pulse oximeter; 2) To assess the agreement between the ring-type wearable device and PSG monitor on OSAS screening.

Study design: Clinical diagnostic trial.

Study population: Individuals who are willing to participate in the study and sign the informed consent are considered to be eligible. Specific inclusion criterias include: 1) Agree to receive overnight polysomnography and wear the ring-type device at the same time; 2) At least 18 years old.

Sample size estimation: About 200 participants.

Timeline: Start of subjects' enrollment: Dec 2022; End of subjects' enrollment: Oct 2023; End of study: Oct 2023.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
Study name: Validation of a Ring-type Wearable Device for Blood Oxygen Monitoring and Obstructive Sleep Apnea Syndrome Screening in Adult Chinese.

Rationale: Obstructive sleep apnoea syndrome (OSAS) is a common chronic sleep-related breathing disorder characterized by repetitive upper airway collapse during sleep, which causes sleep fragmentation, oxygen desaturation, and excessive daytime sleepiness. Previous studies have identified that OSAS is significantly correlated with the risk of cardiovascular and cerebrovascular diseases. Overnight polysomnography (PSG) is the gold standard for diagnosing OSAS at present. However, PSG monitoring requires professional technicists and a lot of channels, which brings inconvenience to both patients and doctors. Wearable devices are growing in popularity and become comfortable, lightweight and technologically advanced for tracking sleep and daily activity.

Objective: 1) To examine the accuracy of blood oxygen monitoring assessed via a ring-type wearable device in comparison to traditional finger clip pulse oximeter; 2) To assess the agreement between the ring-type wearable device and PSG monitor on OSAS screening.

Study design: Clinical diagnostic trial.

Study population: Individuals who are willing to participate in the study and sign the informed consent are considered to be eligible. Specific inclusion criterias include: 1) Agree to receive overnight polysomnography and wear the ring-type device at the same time; 2) At least 18 years old.

Data collections: 1) Data on demographic and clinical characteristics were collected using a questionnaire; 2) Data on blood oxygen saturation and sleep apnea-related parameters were measured by both PSG monitoring and the ring-type wearable device.

Sample size estimation: About 200 participants.

Timeline: Start of subjects' enrollment: Dec 2022; End of subjects' enrollment: Oct 2023; End of study: Oct 2023.

Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

Individuals who are willing to participate in the study and sign the informed consent are considered to be eligible. Specific inclusion criterias include:

1. Agree to receive overnight polysomnography and wear the ring-type device at the same time;
2. At least 18 years old.

Exclusion Criteria:

1. Conditions that influencing overnight polysomnography monitoring, including receiving continuous positive airway pressure treatment and coexisting sleep disorders or insomnia;
2. Participants with cognitive dysfunction who are unable to provide informed consent;
3. Other circumstances that individuals are not appropriate for the study upon the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Difference in the mean oxygen saturation | 1 night

SECONDARY OUTCOMES:
Difference in the lowest oxygen saturation | 1 night
Difference in the apnea-hypopnea index | 1 night
Difference in the oxygen desaturation index | 1 night
Difference in the hypoxic burden | 1 night
Agreement between the ring-type wearable device and PSG monitor on OSAS screening | 1 night
  Sensitivity, specificity, positive predictive value, negative predictive value and area under the ROC curve were used to describe the agreement between the ring-type wearable device and PSG monitor on OSAS screening

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, MD, PhD, Principal Investigator — Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China